CLINICAL TRIAL: NCT01688830
Title: Randomised, Double-blind, Placebo-controlled Phase I Study in Healthy Male Volunteers. to Investigate Safety, Tolerability and Pharmacokinetics of Single Rising Doses of BI 655075 (Part 1) and to Explore the Dose of BI 655075 Effective to Reverse Dabigatran Anticoagulant Activity (Part 2)
Brief Title: Study to Evaluate the Safety, Pharmacokinetics and Pharmacodynamics of BI 655075 Administered Alone or With Dabigatran Etexilate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1321.1; 2012-003611-66 (EudraCT Number: EudraCT)
Record Dates: First submitted 2012-09-17; First posted 2012-09-20 (Estimated); Results first posted 2016-02-15 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-05

CONDITIONS: Healthy
MeSH Terms: interventions — Dabigatran; idarucizumab

ARMS (3):
- BI 655075 (Experimental)
  Interventions: Drug: BI 655075
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- BI 655075 with dabigatran (Experimental)
  Interventions: Drug: Dabigatran; Drug: BI 655075

INTERVENTIONS:
Drug: Dabigatran
  Arms: BI 655075 with dabigatran
Drug: BI 655075
  Arms: BI 655075; BI 655075 with dabigatran
Drug: Placebo
  Arms: Placebo

SUMMARY:
The primary objective is to investigate the safety, tolerability and pharmacokinetics of BI 655075 following intravenous administration of single rising doses of BI 655075 when administered alone and after administration of dabigatran.

ELIGIBILITY:
Inclusion criteria:

1. Healthy male subjects

Exclusion criteria:

1. Any relevant deviation from healthy conditions

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 157 (Actual)
Dates: Start 2012-09; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1321.1.1 Boehringer Ingelheim Investigational Site, Antwerp, Belgium

REFERENCES:
- [Derived] Norris S, Ramael S, Ikushima I, Haazen W, Harada A, Moschetti V, Imazu S, Reilly PA, Lang B, Stangier J, Glund S. Evaluation of the immunogenicity of the dabigatran reversal agent idarucizumab during Phase I studies. Br J Clin Pharmacol. 2017 Aug;83(8):1815-1825. doi: 10.1111/bcp.13269. Epub 2017 Apr 6. PMID 28230262
- [Derived] Glund S, Stangier J, Schmohl M, Gansser D, Norris S, van Ryn J, Lang B, Ramael S, Moschetti V, Gruenenfelder F, Reilly P, Kreuzer J. Safety, tolerability, and efficacy of idarucizumab for the reversal of the anticoagulant effect of dabigatran in healthy male volunteers: a randomised, placebo-controlled, double-blind phase 1 trial. Lancet. 2015 Aug 15;386(9994):680-90. doi: 10.1016/S0140-6736(15)60732-2. Epub 2015 Jun 15. PMID 26088268

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study is conducted in two parts:
  Parts 1 and 2 had a single rising dose design; subjects in Part 3 received 2 single doses 1 h apart.
  Part 1: 8 subjects per dose group Part 2: 12 subjects per dose group Part 3: 12 subjects per dose group
Groups:
- Placebo 1 h: One single intravenous long infusion (1 h) of Idarucizumab Placebo
  This is administered during Part 1 of the study
- 20 mg Idarucizumab 1h: Dose group 1: One single intravenous long infusion (1 h) of 20 mg Idarucizumab verum
  This is administered during Part 1 of the study
- 60 mg Idarucizumab 1h: Dose group 2: One single intravenous long infusion (1 h) of 60 mg Idarucizumab verum
  This is administered during Part 1 of the study
- 200 mg Idarucizumab 1h: Dose group 3: One single intravenous long infusion (1 h) of 200 mg Idarucizumab verum
  This is administered during Part 1 of the study
- 600 mg Idarucizumab 1h: Dose group 4: One single intravenous long infusion (1 h) of 600 mg Idarucizumab verum
  This is administered during Part 1 of the study
- 1.2 g Idarucizumab 1h: Dose group 5: One single intravenous long infusion (1 h) of 1.2 g Idarucizumab verum
  This is administered during Part 1 of the study
- 2 g Idarucizumab 1h: Dose group 6: One single intravenous long infusion (1 h) of 2 g Idarucizumab verum
  This is administered during Part 1 of the study
- 3 g Idarucizumab 1h: Dose group 7: One single intravenous long infusion (1 h) of 3 g Idarucizumab verum
  This is administered during Part 1 of the study
- 4 g Idarucizumab 1h: Dose group 8: One single intravenous long infusion (1 h) of 4 g Idarucizumab verum
  This is administered during Part 1 of the study
- 6 g Idarucizumab 1h: Dose group 9: One single intravenous long infusion (1 h) of 6 g Idarucizumab verum
  This is administered during Part 1 of the study
- 8 g Idarucizumab 1h: Dose group 10: One single intravenous long infusion (1 h) of 8 g Idarucizumab verum
  This is administered during Part 1 of the study
- Placebo 5min: One single intravenous short infusion (5 min) of Idarucizumab Placebo
  This is administered during Part 1 of the study
- 1 g Idarucizumab 5min: Dose group 11: One single intravenous short infusion (5 min) of 1 g Idarucizumab verum
  This is administered during Part 1 of the study
- 2 g Idarucizumab 5min: Dose group 12: One single intravenous short infusion (5 min) of 2 g Idarucizumab verum
  This is administered during Part 1 of the study
- 4 g Idarucizumab 5min: Dose group 13: One single intravenous short infusion (5 min) of 4 g Idarucizumab verum
  This is administered during Part 1 of the study
- DE+ Placebo 5min: One single intravenous short infusion (5 min) of Idarucizumab Placebo administered at or close to the steady state of Dabigatran etexilate (DE) 220 mg.
  This is administered during Part 2 of the study
  DE is administered orally :
  Day 1 to 3: twice daily; Day 4: once daily
- DE+ 1 g Idarucizumab 5min: Dose group 14: One single intravenous short infusion (5 min) of 1 g Idarucizumab verum administered at or close to the steady state of Dabigatran etexilate (DE) 220 mg.
  This is administered during Part 2 of the study.
  DE is administered orally :
  Day 1 to 3: twice daily; Day 4: once daily
- DE+ 2 g Idarucizumab 5min: Dose group 15: One single intravenous short infusion (5 min) of 2 g Idarucizumab verum administered at or close to the steady state of Dabigatran etexilate (DE) 220 mg.
  This is administered during Part 2 of the study.
  DE is administered orally :
  Day 1 to 3: twice daily; Day 4: once daily
- DE+ 4 g Idarucizumab 5min: Dose group 16: One single intravenous short infusion (5 min) of 4 g Idarucizumab verum administered at or close to the steady state of Dabigatran etexilate (DE) 220 mg.
  This is administered during Part 2 of the study.
  DE is administered orally :
  Day 1 to 3: twice daily; Day 4: once daily
- DE+ Placebo+ Placebo: Two short intravenous infusions (5 min each) of Idarucizumab Placebo administered at or close to the steady state of Dabigatran etexilate (DE) 220 mg.
  This is administered during Part 3 of the study
  DE is administered orally :
  Day 1 to 3: twice daily; Day 4: once daily
- DE+ 5 g + 2.5 g Idarucizumab: Dose group 17: Two short intravenous infusions (5 min each) of 7.5 g Idarucizumab verum administered (5 g + 2.5 g 1 h later) at or close to the steady state of Dabigatran etexilate (DE) 220 mg.
  This is administered during Part 3 of the study
  DE is administered orally :
  Day 1 to 3: twice daily; Day 4: once daily
Period: Overall Study
Arm/Group | Placebo 1 h | 20 mg Idarucizumab 1h | 60 mg Idarucizumab 1h | 200 mg Idarucizumab 1h | 600 mg Idarucizumab 1h | 1.2 g Idarucizumab 1h | 2 g Idarucizumab 1h | 3 g Idarucizumab 1h | 4 g Idarucizumab 1h | 6 g Idarucizumab 1h | 8 g Idarucizumab 1h | Placebo 5min | 1 g Idarucizumab 5min | 2 g Idarucizumab 5min | 4 g Idarucizumab 5min | DE+ Placebo 5min | DE+ 1 g Idarucizumab 5min | DE+ 2 g Idarucizumab 5min | DE+ 4 g Idarucizumab 5min | DE+ Placebo+ Placebo | DE+ 5 g + 2.5 g Idarucizumab
Started | 21 | 6 | 6 | 6 | 5 | 6 | 12 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 9 | 9 | 9 | 8 | 3 | 9
Completed | 21 | 6 | 6 | 6 | 5 | 6 | 12 | 6 | 6 | 6 | 5 | 6 | 6 | 6 | 6 | 9 | 9 | 9 | 8 | 3 | 9
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): All randomised subjects who received 1 dose of trial medication were included in the treated set
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo 1 h | 20 mg Idarucizumab 1h | 60 mg Idarucizumab 1h | 200 mg Idarucizumab 1h | 600 mg Idarucizumab 1h | 1.2 g Idarucizumab 1h | 2 g Idarucizumab 1h | 3 g Idarucizumab 1h | 4 g Idarucizumab 1h | 6 g Idarucizumab 1h | 8 g Idarucizumab 1h | Placebo 5min | 1 g Idarucizumab 5min | 2 g Idarucizumab 5min | 4 g Idarucizumab 5min | DE+ Placebo 5min | DE+ 1 g Idarucizumab 5min | DE+ 2 g Idarucizumab 5min | DE+ 4 g Idarucizumab 5min | DE+ Placebo+ Placebo | DE+ 5 g + 2.5 g Idarucizumab | Total
Number analyzed (Participants) | 21 | 6 | 6 | 6 | 5 | 6 | 12 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 9 | 9 | 9 | 8 | 3 | 9 | 157
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.3 (7.8) | 29.8 (6.6) | 35.2 (5.5) | 36.2 (8.8) | 36.6 (4.5) | 32.0 (8.9) | 30.3 (8.5) | 32.7 (4.2) | 35.3 (9.5) | 34.5 (8.8) | 35.2 (9.1) | 34.5 (11.2) | 34.7 (8.5) | 31.8 (5.4) | 36.0 (8.3) | 30.9 (8.9) | 31.3 (7.0) | 31.1 (8.3) | 31.9 (9.1) | 30.0 (2.6) | 29.9 (9.0) | 32.4 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 21 | 6 | 6 | 6 | 5 | 6 | 12 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 9 | 9 | 9 | 8 | 3 | 9 | 157

OUTCOME MEASURES:

1. Secondary Outcome: Cmax (Maximum Measured Concentration) for Idarucizumab
Description: Cmax (maximum measured concentration) for idarucizumab
Time Frame: -2 hours(h), -0.5h, 0h, 2min(m), 5m, 10m, 15m,30m, 45m, 1h, 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 10h, 12h, 16h, 24h, 48h, 72h
Population: Pharmacokinetic set (PKS) comprises of all subjects (with evaluable observations) in the TS who provided at least 1 PK endpoint and had no important protocol violations relevant to the evaluation of PK and additionally for Part 2 and 3 had no emesis with onset at or before twice the median tmax of dabigatran.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | 20 mg Idarucizumab 1h | 60 mg Idarucizumab 1h | 200 mg Idarucizumab 1h | 600 mg Idarucizumab 1h | 1.2 g Idarucizumab 1h | 2 g Idarucizumab 1h | 3 g Idarucizumab 1h | 4 g Idarucizumab 1h | 6 g Idarucizumab 1h | 8 g Idarucizumab 1h | 1 g Idarucizumab 5min | 2 g Idarucizumab 5min | 4 g Idarucizumab 5min | DE+ 1 g Idarucizumab 5min | DE+ 2 g Idarucizumab 5min | DE+ 4 g Idarucizumab 5min | DE+ 5 g + 2.5 g Idarucizumab
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 12 | 6 | 6 | 6 | 5 | 6 | 6 | 6 | 9 | 9 | 8 | 9
nmol/L | 79.9 (15.1) | 257 (11.1) | 809 (13.9) | 2440 (13.1) | 4520 (9.72) | 7420 (15.1) | 11700 (10.4) | 15700 (15.6) | 22100 (12.0) | 33900 (13.2) | 6360 (16.7) | 13600 (23.4) | 21400 (13.1) | 5410 (13.5) | 12500 (21.5) | 25800 (25.1) | 35300 (24.4)

2. Secondary Outcome: Tmax (Time From Dosing to Maximum Measured Concentration) for Idarucizumab
Description: tmax (time from dosing to maximum measured concentration) for idarucizumab
Time Frame: as for outcome 1
Population: PKS (presented values are those subjects from the PKS with evaluable observations for this endpoint)
Measure: Median (Full Range); unit: hours
Arm/Group | 20 mg Idarucizumab 1h | 60 mg Idarucizumab 1h | 200 mg Idarucizumab 1h | 600 mg Idarucizumab 1h | 1.2 g Idarucizumab 1h | 2 g Idarucizumab 1h | 3 g Idarucizumab 1h | 4 g Idarucizumab 1h | 6 g Idarucizumab 1h | 8 g Idarucizumab 1h | 1 g Idarucizumab 5min | 2 g Idarucizumab 5min | 4 g Idarucizumab 5min | DE+ 1 g Idarucizumab 5min | DE+ 2 g Idarucizumab 5min | DE+ 4 g Idarucizumab 5min | DE+ 5 g + 2.5 g Idarucizumab
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 12 | 6 | 6 | 6 | 5 | 6 | 6 | 6 | 9 | 9 | 8 | 9
hours | 1.00 [0.967 to 1.17] | 1.03 [0.967 to 1.17] | 1.03 [0.967 to 1.08] | 1.10 [1.03 to 1.18] | 0.967 [0.967 to 1.08] | 0.984 [0.967 to 1.17] | 1.00 [0.967 to 1.05] | 1.06 [0.967 to 1.17] | 1.03 [0.967 to 1.08] | 1.08 [0.967 to 1.17] | 0.117 [0.0830 to 0.167] | 0.142 [0.117 to 0.250] | 0.167 [0.117 to 0.250] | 0.117 [0.0830 to 0.167] | 0.200 [0.167 to 0.333] | 0.117 [0.0830 to 0.167] | 0.117 [0.0830 to 1.12]

3. Secondary Outcome: AUC0-inf (Area Under the Concentration-time Curve From Time 0 Extrapolated to Infinity) for Idarucizumab
Description: AUC0-inf (area under the concentration-time curve from time 0 extrapolated to infinity) for idarucizumab
Time Frame: as for outcome 1
Population: PKS (presented values are those subjects from the PKS with evaluable observations for this endpoint)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | 20 mg Idarucizumab 1h | 60 mg Idarucizumab 1h | 200 mg Idarucizumab 1h | 600 mg Idarucizumab 1h | 1.2 g Idarucizumab 1h | 2 g Idarucizumab 1h | 3 g Idarucizumab 1h | 4 g Idarucizumab 1h | 6 g Idarucizumab 1h | 8 g Idarucizumab 1h | 1 g Idarucizumab 5min | 2 g Idarucizumab 5min | 4 g Idarucizumab 5min | DE+ 1 g Idarucizumab 5min | DE+ 2 g Idarucizumab 5min | DE+ 4 g Idarucizumab 5min | DE+ 5 g + 2.5 g Idarucizumab
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 12 | 6 | 6 | 6 | 5 | 6 | 6 | 6 | 9 | 9 | 8 | 9
nmol*h/L | 146 (19.8) | 426 (11.6) | 1950 (129) | 6970 (75.4) | 8780 (4.92) | 14500 (15.9) | 22600 (17.6) | 31000 (12.9) | 41200 (11.8) | 63800 (15.6) | 7790 (13.1) | 16400 (16.8) | 25800 (22.1) | 6480 (17.1) | 16600 (10.7) | 30900 (14.1) | 62300 (8.43)

4. Secondary Outcome: Aet1-t2 (Amount of Idarucizumab Eliminated in Urine From Time Point t1 to Time Point t2)
Description: Aet1-t2 (amount of idarucizumab eliminated in urine from time point t1 to time point t2)
  Ae(0-7h) is presented for dose groups with 1 h infusion and Ae(0-4h) is presented for dose groups with 5 min infusion.
Time Frame: Up to 7 hours
Population: PKS (presented values are those subjects from the PKS with evaluable observations for this endpoint)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μmol
Arm/Group | 20 mg Idarucizumab 1h | 60 mg Idarucizumab 1h | 200 mg Idarucizumab 1h | 600 mg Idarucizumab 1h | 1.2 g Idarucizumab 1h | 2 g Idarucizumab 1h | 3 g Idarucizumab 1h | 4 g Idarucizumab 1h | 6 g Idarucizumab 1h | 8 g Idarucizumab 1h | 1 g Idarucizumab 5min | 2 g Idarucizumab 5min | 4 g Idarucizumab 5min | DE+ 1 g Idarucizumab 5min | DE+ 2 g Idarucizumab 5min | DE+ 4 g Idarucizumab 5min | DE+ 5 g + 2.5 g Idarucizumab
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 6 | 12 | 6 | 6 | 6 | 5 | 6 | 6 | 6 | 9 | 9 | 8 | 9
μmol | NA (NA) — Missing values (denoted with 'NA') were not measured for the respective dose groups. | NA (NA) — Missing values (denoted with 'NA') were not measured for the respective dose groups. | NA (NA) — Missing values (denoted with 'NA') were not measured for the respective dose groups. | NA (NA) — Missing values (denoted with 'NA') were not measured for the respective dose groups. | NA (NA) — Missing values (denoted with 'NA') were not measured for the respective dose groups. | NA (NA) — Missing values (denoted with 'NA') were not measured for the respective dose groups. | NA (NA) — Missing values (denoted with 'NA') were not measured for the respective dose groups. | NA (NA) — Missing values (denoted with 'NA') were not measured for the respective dose groups. | 36.1 (50.1) | 39.5 (395) | 2.23 (76.3) | 8.00 (73.1) | 32.6 (23.6) | 1.71 (90.6) | 11.0 (23.4) | 33.6 (30.5) | 73.5 (24.9)

5. Primary Outcome: Number of Subjects With Drug Related Adverse Events (AE)
Description: Frequency of subjects with related adverse events (AE) by treatment
Time Frame: AEs occurring until end of follow-up (Up to 3 months after last drug administration)
Population: Treated set
Measure: Number; unit: participants
Arm/Group | Placebo 1 h | 20 mg Idarucizumab 1h | 60 mg Idarucizumab 1h | 200 mg Idarucizumab 1h | 600 mg Idarucizumab 1h | 1.2 g Idarucizumab 1h | 2 g Idarucizumab 1h | 3 g Idarucizumab 1h | 4 g Idarucizumab 1h | 6 g Idarucizumab 1h | 8 g Idarucizumab 1h | Placebo 5min | 1 g Idarucizumab 5min | 2 g Idarucizumab 5min | 4 g Idarucizumab 5min | DE+ Placebo 5min | DE+ 1 g Idarucizumab 5min | DE+ 2 g Idarucizumab 5min | DE+ 4 g Idarucizumab 5min | DE+ Placebo+ Placebo | DE+ 5 g + 2.5 g Idarucizumab
Number analyzed (Participants) | 21 | 6 | 6 | 6 | 5 | 6 | 12 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 9 | 9 | 9 | 8 | 3 | 9
participants | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1

6. Secondary Outcome: Aet1-t2,ss (Amount of Dabigatran Etexilate Eliminated in Urine From Time Point t1 to Time Point t2, at Steady State) on Day 3 and Day 4 for Sum Dabigatran
Description: Aet1-t2,ss (amount of dabigatran etexilate eliminated in urine from time point t1 to time point t2, at steady state) on Day 3 and Day 4
  Ae(0-12h,ss) of sum dabigatran
Time Frame: Intervals 0-2, 2-6, 6-10, 10-12 hours on Day 3 post dabigatran treatment and -2 to -0:05, -0:05 to 4, 4-8, 8-10, 10-12, 12-24, 24-48, 48-72 on Day 4 post Idarucizumab treatment
Population: PKS (presented values are those subjects from the PKS with evaluable observations for this endpoint)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg
Groups:
- DE (Dose Groups 14-16: Day 3): Dabigatran etexilate (220 mg; 2 capsules, each 110 mg) was administered to subjects orally, both in the mornings and evenings of Days 1 to 3 in dose groups 14-16
- DE+ 1 g Idarucizumab 5min: One single intravenous short infusion (5 min) of 1 g Idarucizumab verum administered at or close to the steady state of Dabigatran etexilate (DE) 220 mg.
  This is administered during Part 2 of the study.
  DE is administered orally :
  Day 1 to 3: twice daily; Day 4: once daily
- DE+ 2 g Idarucizumab 5min; DE+ 4 g Idarucizumab 5min: One single intravenous short infusion (5 min) of 2 g Idarucizumab verum administered at or close to the steady state of Dabigatran etexilate (DE) 220 mg.
  This is administered during Part 2 of the study.
  DE is administered orally :
  Day 1 to 3: twice daily; Day 4: once daily
- DE (Dose Groups 17: Day 3): Dabigatran etexilate (220 mg; 2 capsules, each 110 mg) was administered to subjects orally, both in the mornings and evenings of Days 1 to 3 in dose group 17
Arm/Group | DE (Dose Groups 14-16: Day 3) | DE+ Placebo 5min | DE+ 1 g Idarucizumab 5min | DE+ 2 g Idarucizumab 5min | DE+ 4 g Idarucizumab 5min | DE (Dose Groups 17: Day 3) | DE+ Placebo+ Placebo | DE+ 5 g + 2.5 g Idarucizumab
Number analyzed (Participants) | 34 | 9 | 9 | 9 | 8 | 12 | 2 | 8
μg | 6600 (54.4) | 6870 (37.8) | 5160 (57.1) | 3820 (86.9) | 3860 (39.1) | 6420 (38.7) | 5060 (55.1) | 4290 (35.2)

7. Secondary Outcome: C1.92,ss, C2,ss, C2.5,ss, C6,ss, and C12,ss (Concentration of the Unbound Sum Dabigatran in Plasma at Steady State)
Description: Concentrations of unbound sum dabigatran in plasma after 1.92 to 12 h, at steady state of dabigatran, on Day 4 are presented.
  The endpoint refers to unbound sum dabigatran at several time points. The intended pharmacodynamic effect of idarucizumab is to reduce the concentration of this measure to levels below the lower limit of quantification (BLQ). "BLQ" values are not considered in the calculation of descriptive statistics; and therefore bias the result. This is the reason for applying the 2/3 rule to obtain reliable results. 2/3 rule states that, Statistics of PK parameters are only estimated when at least 2/3 of the data are evaluable.
Time Frame: 1.92 hours (h), 2 h, 2.5 h, 6 h and 12 h on Day 4
Population: Pharmadynamic set (PDS) : The PDS was used for all PD analyses and comprised all subjects in the TS who provided at least 1 evaluable predose and
  1 on-treatment observation for calculating ratio (PD endpoint) and who had no important protocol violations relevant to the evaluation of PD.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | DE+ Placebo 5min | DE+ 1 g Idarucizumab 5min | DE+ 2 g Idarucizumab 5min | DE+ 4 g Idarucizumab 5min | DE+ Placebo+ Placebo | DE+ 5 g + 2.5 g Idarucizumab
Number analyzed (Participants) | 9 | 9 | 9 | 8 | 2 | 8
ng/mL
  C1.92,ss (N= 9, 9, 9, 8, 2, 8) | 119 (38.0) | 136 (51.8) | 96.2 (33.3) | 135 (47.6) | 101 (97.8) | 112 (34.0)
  C2,ss (N= 9, 6, NA, NA, 2, NA) | 123 (40.8) | 1.59 (10.7) | NA (NA) — NA: Not calculated, reliable estimation can only be performed when at least 2/3 of the data are available and thus not calculated according to internal rules | NA (NA) — NA: Not calculated, reliable estimation can only be performed when at least 2/3 of the data are available and thus not calculated according to internal rules | 95.6 (109) | NA (NA) — NA: Not calculated, reliable estimation can only be performed when at least 2/3 of the data are available and thus not calculated according to internal rules
  C2.5,ss (N= 9, NA, NA, NA, 2, NA ) | 130 (47.9) | NA (NA) — NA: Not calculated, reliable estimation can only be performed when at least 2/3 of the data are available and thus not calculated according to internal rules | NA (NA) — NA: Not calculated, reliable estimation can only be performed when at least 2/3 of the data are available and thus not calculated according to internal rules | NA (NA) — NA: Not calculated, reliable estimation can only be performed when at least 2/3 of the data are available and thus not calculated according to internal rules | 92.9 (99.4) | NA (NA) — NA: Not calculated, reliable estimation can only be performed when at least 2/3 of the data are available and thus not calculated according to internal rules
  C6,ss (N= 9, 9, NA, NA, 2, NA) | 79.2 (44.6) | 15.3 (296) | NA (NA) — NA: Not calculated, reliable estimation can only be performed when at least 2/3 of the data are available and thus not calculated according to internal rules | NA (NA) — NA: Not calculated, reliable estimation can only be performed when at least 2/3 of the data are available and thus not calculated according to internal rules | 54.8 (93.2) | NA (NA) — NA: Not calculated, reliable estimation can only be performed when at least 2/3 of the data are available and thus not calculated according to internal rules
  C12,ss (N= 9, 9, NA, NA, 2, NA) | 38.5 (40.3) | 18.2 (71.1) | NA (NA) — NA: Not calculated, reliable estimation can only be performed when at least 2/3 of the data are available and thus not calculated according to internal rules | NA (NA) — NA: Not calculated, reliable estimation can only be performed when at least 2/3 of the data are available and thus not calculated according to internal rules | 28.9 (90.6) | NA (NA) — NA: Not calculated, reliable estimation can only be performed when at least 2/3 of the data are available and thus not calculated according to internal rules

8. Secondary Outcome: AUCt1-t2,ss (Area Under the Concentration-time Curve for the Unbound Sum Dabigatran in Plasma From Time Point t1 to Time Point t2, at Steady State) on Day 3 and Day 4
Description: AUC(2-12),ss ((area under the concentration-time curve for the idarucizumab in plasma from time point 2 to 12 h )) on Day 3 and Day 4
Time Frame: 2h, 2.5h, 3h, 4h, 6h, 8h, 10h, 12h
Population: PKS (presented values are those subjects from the PKS with evaluable observations for this endpoint)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | DE (Dose Groups 14-16: Day 3) | DE+ Placebo 5min | DE+ 1 g Idarucizumab 5min | DE+ 2 g Idarucizumab 5min | DE+ 4 g Idarucizumab 5min | DE (Dose Groups 17: Day 3) | DE+ Placebo+ Placebo | DE+ 5 g + 2.5 g Idarucizumab
Number analyzed (Participants) | 35 | 9 | 9 | 9 | 8 | 12 | 2 | 8
ng*h/mL | 805 (57.4) | 754 (45.6) | 161 (148) | 20.9 (199) | 11.9 (44.3) | 786 (40.1) | 542 (98.9) | 10.0 (0.344)

9. Secondary Outcome: AUECt1-t2 (Area Under the Effect Curve From Time Point t1 to Time Point t2) on Day 3 and Day 4 (Determined Under Consideration of the Baseline Value) for Part 2 of the Study
Description: AUECt1-t2 (area under the effect curve from time point t1=2 hours to time point t2=12 hours) on Day 3 and Day 4 (determined under consideration of the baseline value).
  Ratio of above baseline AUEC(2-12) on Day 4 to above baseline AUEC(2-12) on Day 3 is presented.
  This endpoint was determined for Activated Partial Thromboplastin time (aPTT), Dithiothreitol (dTT), Thrombin time (TT) and Ecarin clotting time (ECT)
Time Frame: 2hours-12 hours
Population: Pharmacodynamic set (PDS) : The PDS was used for all PD analyses and comprised all subjects in the TS who provided at least 1 evaluable predose and
  1 on-treatment observation for calculating ratio (PD endpoint) and who had no important protocol violations relevant to the evaluation of PD.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | DE+ Placebo 5min | DE+ 1 g Idarucizumab 5min | DE+ 2 g Idarucizumab 5min | DE+ 4 g Idarucizumab 5min
Number analyzed (Participants) | 9 | 9 | 9 | 8
ratio
  aPTT | 1.28 (0.399) | 0.46 (0.342) | 0.14 (0.135) | 0.07 (0.103)
  dTT | 1.01 (0.484) | 0.26 (0.245) | 0.06 (0.094) | 0.02 (0.016)
  TT | 1.08 (0.361) | 0.32 (0.280) | 0.06 (0.124) | 0.00 (0.007)
  ECT | 1.04 (0.493) | 0.28 (0.231) | 0.07 (0.080) | 0.03 (0.013)

10. Secondary Outcome: AUECt1-t2 (Area Under the Effect Curve From Time Point t1 to Time Point t2) on Day 3 and Day 4 (Determined Under Consideration of the Baseline Value) for Part 3 of the Study
Description: AUECt1-t2 (area under the effect curve from time point t1=2 hours to time point t2=12 hours) on Day 3 and Day 4 (determined under consideration of the baseline value).
  Ratio of above baseline AUEC(2-12) on Day 4 to above baseline AUEC(2-12) on Day 3 is presented.
  This endpoint was determined for Activated Partial Thromboplastin time (aPTT) and Dithiothreitol (dTT)
Time Frame: 2hours-12 hours
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | DE+ Placebo+ Placebo | DE+ 5 g + 2.5 g Idarucizumab
Number analyzed (Participants) | 3 | 9
ratio
  aPTT | 1.68 (0.534) | 0.03 (0.045)
  dTT | 1.02 (1.036) | 0.01 (0.029)

ADVERSE EVENTS:
Time Frame: AEs occurring until end of follow-up (Up to 3 months after last drug administration)
Description: AEs occurring between first administration of BI 655075 (5g) and second administration of BI 655075 2.5g are presented separately (shown under "DE + 5g"), and AEs occurring between second administration of BI 655075 2.5g and date of day after trial completion at 0:00h from this group of subjects are presented separately shown under DE+5g+2.5g.
Groups:
- Placebo 1 h: One single intravenous long infusion (1 h) of Idarucizumab Placebo
- 20 mg Idarucizumab 1h: One single intravenous long infusion (1 h) of 20 mg Idarucizumab verum
- 60 mg Idarucizumab 1h: One single intravenous long infusion (1 h) of 60 mg Idarucizumab verum
- 200 mg Idarucizumab 1h: One single intravenous long infusion (1 h) of 200 mg Idarucizumab verum
- 600 mg Idarucizumab 1h: One single intravenous long infusion (1 h) of 600 mg Idarucizumab verum
- 1.2 g Idarucizumab 1h: One single intravenous long infusion (1 h) of 1.2 g Idarucizumab verum
- 2 g Idarucizumab 1h: One single intravenous long infusion (1 h) of 2 g Idarucizumab verum
- 3 g Idarucizumab 1h: One single intravenous long infusion (1 h) of 3 g Idarucizumab verum
- 4 g Idarucizumab 1h: One single intravenous long infusion (1 h) of 4 g Idarucizumab verum
- 6 g Idarucizumab 1h: One single intravenous long infusion (1 h) of 6 g Idarucizumab verum
- 8 g Idarucizumab 1h: One single intravenous long infusion (1 h) of 8 g Idarucizumab verum
- Placebo 5min: One single intravenous short infusion (5 min) of Idarucizumab Placebo
- 1 g Idarucizumab 5min: One single intravenous short infusion (5 min) of 1 g Idarucizumab verum
- 2 g Idarucizumab 5min: Dose group 12: One single intravenous short infusion (5 min) of 2 g Idarucizumab verum
- 4 g Idarucizumab 5min: One single intravenous short infusion (5 min) of 4 g Idarucizumab verum
- DE (Dose Groups 14-16): Dabigatran etexilate (220 mg; 2 capsules, each 110 mg) was administered to subjects orally, both in the mornings and evenings of Days 1 to 3 and in the morning of Day 4 in dose groups 14-16
- DE+ Placebo 5min; DE+ Placebo: One single intravenous short infusion (5 min) of Idarucizumab Placebo administered at or close to the steady state of Dabigatran etexilate (DE) 220 mg.
  DE is administered orally :
  Day 1 to 3: twice daily; Day 4: once daily
- DE+ 1 g Idarucizumab 5min: One single intravenous short infusion (5 min) of 1g of Idarucizumab verum administered at or close to the steady state of Dabigatran etexilate (DE) 220 mg.
  DE is administered orally :
  Day 1 to 3: twice daily; Day 4: once daily
- DE+ 4 g Idarucizumab 5min: One single intravenous short infusion (5 min) of 4 g Idarucizumab verum administered at or close to the steady state of Dabigatran etexilate (DE) 220 mg.
  DE is administered orally :
  Day 1 to 3: twice daily; Day 4: once daily
- DE+ 2 g Idarucizumab 5min: One single intravenous short infusion (5 min) of 2 g Idarucizumab verum administered at or close to the steady state of Dabigatran etexilate (DE) 220 mg.
  DE is administered orally :
  Day 1 to 3: twice daily; Day 4: once daily
- DE (Dose Groups 17): Dabigatran etexilate (220 mg; 2 capsules, each 110 mg) was administered to subjects orally, both in the mornings and evenings of Days 1 to 3 and in the morning of Day 4 in dose group 17
- DE+ Placebo+ Placebo: Two short intravenous infusions (5 min each) of Idarucizumab Placebo administered at or close to the steady state of Dabigatran etexilate (DE) 220 mg.
  DE is administered orally :
  Day 1 to 3: twice daily; Day 4: once daily
- DE+ 5 g: One single intravenous short infusion (5 min) of 5 g Idarucizumab verum administered at or close to the steady state of Dabigatran etexilate (DE) 220 mg.
  DE is administered orally :
  Day 1 to 3: twice daily; Day 4: once daily
- DE+ 5 g + 2.5 g Idarucizumab: Two short intravenous infusions (5 min each) of 7.5 g Idarucizumab verum administered (5 g + 2.5 g 1 h later) at or close to the steady state of Dabigatran etexilate (DE) 220 mg.
  DE is administered orally :
  Day 1 to 3: twice daily; Day 4: once daily
Arm/Group | Placebo 1 h | 20 mg Idarucizumab 1h | 60 mg Idarucizumab 1h | 200 mg Idarucizumab 1h | 600 mg Idarucizumab 1h | 1.2 g Idarucizumab 1h | 2 g Idarucizumab 1h | 3 g Idarucizumab 1h | 4 g Idarucizumab 1h | 6 g Idarucizumab 1h | 8 g Idarucizumab 1h | Placebo 5min | 1 g Idarucizumab 5min | 2 g Idarucizumab 5min | 4 g Idarucizumab 5min | DE (Dose Groups 14-16) | DE+ Placebo 5min | DE+ 1 g Idarucizumab 5min | DE+ 4 g Idarucizumab 5min | DE+ 2 g Idarucizumab 5min | DE (Dose Groups 17) | DE+ Placebo | DE+ Placebo+ Placebo | DE+ 5 g | DE+ 5 g + 2.5 g Idarucizumab
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/6 | 0/6 | 0/6 | 0/5 | 0/6 | 0/12 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/35 | 0/9 | 0/9 | 0/8 | 0/9 | 0/12 | 0/3 | 0/3 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 7/21 | 2/6 | 2/6 | 5/6 | 2/5 | 1/6 | 4/12 | 3/6 | 0/6 | 1/6 | 2/6 | 2/6 | 3/6 | 2/6 | 3/6 | 20/35 | 1/9 | 4/9 | 4/8 | 4/9 | 2/12 | 0/3 | 1/3 | 1/9 | 3/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo 1 h (N=21) | 20 mg Idarucizumab 1h (N=6) | 60 mg Idarucizumab 1h (N=6) | 200 mg Idarucizumab 1h (N=6) | 600 mg Idarucizumab 1h (N=5) | 1.2 g Idarucizumab 1h (N=6) | 2 g Idarucizumab 1h (N=12) | 3 g Idarucizumab 1h (N=6) | 4 g Idarucizumab 1h (N=6) | 6 g Idarucizumab 1h (N=6) | 8 g Idarucizumab 1h (N=6) | Placebo 5min (N=6) | 1 g Idarucizumab 5min (N=6) | 2 g Idarucizumab 5min (N=6) | 4 g Idarucizumab 5min (N=6) | DE (Dose Groups 14-16) (N=35) | DE+ Placebo 5min (N=9) | DE+ 1 g Idarucizumab 5min (N=9) | DE+ 4 g Idarucizumab 5min (N=8) | DE+ 2 g Idarucizumab 5min (N=9) | DE (Dose Groups 17) (N=12) | DE+ Placebo (N=3) | DE+ Placebo+ Placebo (N=3) | DE+ 5 g (N=9) | DE+ 5 g + 2.5 g Idarucizumab (N=9)
Nasopharyngitis (Infections and infestations) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 1 | 0 | 2 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 3 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Skin reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Glycosuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Catheter site pain (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Feeling hot (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Infusion site swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site haematoma (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Application site irritation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
There is only one group of subjects in study part 3 receiving active treatment. However, AE table displays the AEs occurring in different phases separately.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights